CLINICAL TRIAL: NCT00129220
Title: Placebo- and Haloperidol-Controlled Double-Blind Trial of Olanzapine in Patients With Manic or Mixed Episode of Bipolar I Disorder
Brief Title: Trial of Olanzapine in Patients With Manic or Mixed Episode of Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9636; F1D-JE-BMAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-08-08; First posted 2005-08-11 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Bipolar Disorder
Keywords: Manic or mixed episode associated with bipolar I disorder
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Olanzapine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Olanzapine (Experimental): olanzapine: 5 to 20 mg per day for 6 weeks
  Interventions: Drug: olanzapine
- Haloperidol (Active Comparator): haloperidol: 2.5 to 10 mg per day for 6 weeks
  Interventions: Drug: haloperidol
- Placebo (Placebo Comparator): placebo for 3 weeks, then olanzapine 5 to 20 mg per day for 3 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: olanzapine — 5-20 mg, oral, once daily (evening), for 6 weeks
  Other Names: LY170053; Zyprexa
  Arms: Olanzapine
Drug: haloperidol — 2.5-10 mg, oral, twice daily (morning and evening), for 6 weeks.
  Arms: Haloperidol
Drug: placebo — placebo, oral tablets, twice daily (morning and evening), for 3 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm the efficacy of olanzapine in the treatment of manic or mixed symptoms associated with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for manic or mixed episodes according to the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) and have a diagnosis of "294.4x Bipolar I Disorder, Most Recent Episode Manic" or "296.6x Bipolar I Disorder, Most Recent Episode Mixed".
* Have a total score on the Young Mania Rating Scale (YMRS) of at least 20 at Visit 1 and Visit 2.

Exclusion Criteria:

* Have received an antidepressant or a psychostimulant within 5 days prior to Visit 1.
* The duration of the current episode is more than 90 days at Visit 1.
* Have a history or a diagnosis of diabetes mellitus.
* Have received any psychotropic medication within 2 days prior to Visit 2 (except for benzodiazepines).

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2005-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Monday-Friday 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Japan (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okinawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

REFERENCES:
- [Derived] Katagiri H, Takita Y, Tohen M, Higuchi T, Kanba S, Takahashi M. Efficacy and safety of olanzapine in the treatment of Japanese patients with bipolar I disorder in a current manic or mixed episode: a randomized, double-blind, placebo- and haloperidol-controlled study. J Affect Disord. 2012 Feb;136(3):476-84. doi: 10.1016/j.jad.2011.10.045. Epub 2011 Nov 30. PMID 22134043

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period I was a week-long Screening Period. Study Period II was a 3-week-long Early Double-Blind Period. Study Period III was a 3-week-long Last Double-Blind Period.
Period: Study Period II
Arm/Group | Olanzapine | Haloperidol | Placebo
Started | 105 | 20 | 99
Received at Least One Dose of Study Drug | 104 | 20 | 97
Completed | 72 | 8 | 52
Not Completed | 33 | 12 | 47
Not completed — Adverse Event | 9 | 5 | 7
Not completed — Lack of Efficacy | 15 | 1 | 28
Not completed — Entry Criteria Not Met | 2 | 0 | 2
Not completed — Protocol Violation | 4 | 2 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 4
Not completed — Reason Not Specified | 2 | 0 | 5
Period: Study Period III
Arm/Group | Olanzapine | Haloperidol | Placebo
Started | 72 | 8 | 52
Completed | 59 | 7 | 42
Not Completed | 13 | 1 | 10
Not completed — Adverse Event | 1 | 0 | 3
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Reason Not Specified | 9 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Haloperidol | Placebo | Total
Number analyzed (Participants) | 104 | 20 | 97 | 221
Age Continuous [Mean (Standard Deviation); unit: years] | 43.1 (12.0) | 49.3 (11.9) | 42.5 (10.9) | 43.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 9 | 57 | 121
  Male | 49 | 11 | 40 | 100
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 104 | 20 | 97 | 221
Region of Enrollment [Number; unit: participants]
  Japan | 104 | 20 | 97 | 221
Current Illness Episode: Manic versus Mixed [Number; unit: participants]
  Manic | 95 | 19 | 89 | 203
  Mixed | 9 | 1 | 8 | 18
Current Illness Episode: Psychotic versus Nonpsychotic [Number; unit: participants]
  Psychotic | 17 | 4 | 19 | 40
  Nonpsychotic | 87 | 16 | 78 | 181
Hospitalization Status [Number; unit: participants]
  In-Patients | 41 | 10 | 38 | 89
  Out-Patients | 63 | 10 | 59 | 132
Psychosis [Number; unit: participants] — Type of psychosis for those participants who had a current illness episode of psychotic (total number of participants with data in this baseline measure will be less than the total in each arm)
  participants
    Mood-Congruent | 16 | 4 | 19 | 39
    Mood-Incongruent | 1 | 0 | 0 | 1
17-Item Hamilton Depression Rating Scale Total Score [Mean (Standard Deviation); unit: units on a scale] — The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
  units on a scale | 4.5 (3.9) | 4.1 (3.7) | 4.9 (4.5) | 4.7 (4.1)
Age of Onset of Illness [Mean (Standard Deviation); unit: years] | 31.2 (11.6) | 37.7 (12.5) | 30.9 (10.7) | 31.6 (11.4)
Clinical Global Impression-Severity of Illness, Bipolar Version (CGI-BP) [Mean (Standard Deviation); unit: units on a scale] — A global rating scale for severity of patients adapted to bipolar disorder. Measures severity of the patient's overall severity of manic symptoms, depressive symptoms, and overall mood symptoms. Each of the three symptoms are on a scale of 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale
    Mania | 4.2 (1.0) | 4.6 (0.8) | 4.1 (1.1) | 4.2 (1.0)
    Depression | 1.3 (0.6) | 1.1 (0.2) | 1.3 (0.7) | 1.2 (0.6)
    Overall Mood | 4.1 (1.0) | 4.4 (1.2) | 4.1 (1.1) | 4.1 (1.1)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 162.74 (8.07) | 162.10 (7.87) | 163.09 (9.66) | 162.84 (8.76)
Length of Current Illness Episode [Mean (Standard Deviation); unit: days] | 34.6 (22.9) | 34.2 (22.0) | 33.5 (25.4) | 34.1 (23.9)
Positive and Negative Syndrome Scale Positive Subscale Score [Mean (Standard Deviation); unit: units on a scale] — Assesses positive symptoms associated with schizophrenia. 7 items make up the Positive scale (ex. delusions, conceptual disorganization, and hallucinatory behavior). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total Positive Subscale scores range from 7 to 49. For this study, the score was converted to 0 to 6 for each item range; hence, the total positive subscale score ranges from 0 to 42.
  units on a scale | 11.5 (4.8) | 11.3 (4.5) | 10.7 (4.7) | 11.1 (4.7)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 60.88 (11.69) | 59.20 (9.87) | 61.86 (13.78) | 61.17 (12.49)
Young Mania Rating Scale (YMRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
  units on a scale | 27.7 (5.9) | 26.6 (4.5) | 26.9 (5.6) | 27.3 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 3 Week Endpoint in Young Mania Rating Scale (YMRS) Total Score
Description: The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: Baseline, 3 weeks
Population: Participants in the Full Analysis Set: participants who had baseline and post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 104 | 20 | 97
units on a scale | -12.6 (10.0) | -14.3 (11.4) | -6.8 (14.0)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Squares Mean Difference = -5.62, 95% CI 2-sided [-8.87 to -2.37] — Least Squares Mean Difference = Olanzapine minus Placebo

2. Secondary Outcome: Change From Baseline to 6 Week Endpoint in Young Mania Rating Scale (YMRS)
Description: as for outcome 1
Time Frame: Baseline, 6 weeks
Population: Participants in the Full Analysis Set: participants who had baseline and post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 104 | 20 | 97
units on a scale | -16.0 (11.4) | -14.7 (13.1) | -10.1 (15.8)
Statistical Analysis 1: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.774, ANCOVA; Least Squares Mean Difference = -0.78, 95% CI 2-sided [-6.15 to 4.59] — Least Squares Mean Difference = Olazapine minus Haloperidol

3. Secondary Outcome: Remission Rate of Bipolar Disorder (Olanzapine Versus Haloperidol)
Description: Remission of bipolar disorder was defined as completing the 6-week period with meeting the criteria for Young Mania Rating Scale (YMRS) total score of 12 or less and 17-Item Hamilton Depression Rating Scale (HAMD-17) total scores of 7 or less at Week 6. YMRS is an 11-item scale measuring severity of manic episodes; total score ranges = 0 (normal) to 60 (severe). The 17-item HAMD measures depression severity; total score ranges = 0 (normal) to 52 (severe). Remission Rate (percent) = number of patients meeting remission criteria divided by number of patients in treatment arm, multiplied by 100.
Time Frame: 6 weeks
Population: Participants in the Full Analysis Set: participants who had baseline and post-baseline measurement.
Measure: Number; unit: percentage of participants
Groups:
- Olanzapine: olanzapine: 5 to 20 mg per day
- Haloperidol: haloperidol: 2.5 to 10 mg per day
Arm/Group | Olanzapine | Haloperidol
Number analyzed (Participants) | 104 | 20
percentage of participants | 44.2 | 20.0
Statistical Analysis 1: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.064, Cochran-Mantel-Haenszel; Least Squares Mean Difference = 21.0, 95% CI 2-sided [1.6 to 40.4] — Least Squares Mean Difference = Olanzapine minus Haloperidol

4. Secondary Outcome: Change From Baseline to 6 Week Endpoint in Clinical Global Impressions - Bipolar Version (CGI-BP), Overall Severity of Illness
Description: A global rating scale for severity of patients adapted to bipolar disorder. Measures severity of the patient's overall severity of overall mood symptoms on a scale of 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, 6 weeks
Population: Participants in the Full Analysis Set: participants who had baseline and post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 104 | 20 | 97
units on a scale | -1.6 (1.5) | -1.3 (1.8) | -0.9 (1.7)
Statistical Analysis 1: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.171, ANCOVA; Least Squares Mean Difference = -0.47, 95% CI 2-sided [-1.15 to 0.21] — Least Squares Mean Difference = Olanzapine minus Haloperidol

5. Secondary Outcome: Change From Baseline to 3 Week and 6 Week Endpoints in Clinical Global Impression - Bipolar Version (CGI-BP) Mania Subscale
Description: A global rating scale for severity of patients adapted to bipolar disorder. Measures severity of the patient's overall severity of manic symptoms on a scale of 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, 3 weeks, 6 weeks
Population: Participants in the Full Analysis Set: participants who had baseline and post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 104 | 20 | 97
units on a scale
  3-Week Change | -1.2 (1.2) | -1.7 (1.7) | -0.6 (1.5)
  6-Week Change | -1.7 (1.5) | -1.9 (1.9) | -1.0 (1.7)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value for 3-Week Change; Least Squares Mean Difference = -0.51, 95% CI 2-sided [-0.87 to -0.15] — Least Squares Mean Difference = Olanzapine minus Placebo
Statistical Analysis 2: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.722, ANCOVA — P-value for 6-Week Change; Least Squares Mean Difference = -0.13, 95% CI 2-sided [-0.82 to 0.57] — Least Squares Mean Difference = Olanzapine minus Haloperidol

6. Secondary Outcome: Response Rate of Manic Symptoms at 3 Weeks and 6 Weeks
Description: Participants who had 50 percent or more decrease from the baseline in YMRS total scores were defined as a responder. The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60. Response Rate (percent) = number of patients meeting response criterion for manic symptom divided by number of patients in treatment arm, multiplied by 100.
Time Frame: Baseline, 3 weeks, 6 weeks
Population: Participants in the Full Analysis Set: participants who had baseline and post-baseline measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 104 | 20 | 97
percentage of participants
  3 Week Response Rate | 51.0 | 65.0 | 44.3
  6 Week Response Rate | 67.3 | 65.0 | 55.7
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.333, Cochran-Mantel-Haenszel — P-value for 3-Week Response Rate; Mean Difference (Net) = 6.7, 95% CI 2-sided [-6.7 to 20.1]
Statistical Analysis 2: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.908, Cochran-Mantel-Haenszel — P-value for 6-Week Response Rate; Mean Difference (Net) = -1.3, 95% CI 2-sided [-21.0 to 18.4]

7. Secondary Outcome: Remission Rate of Manic Symptoms at 3 Weeks and 6 Weeks
Description: Participants who had a YMRS total score of 12 or less were considered to be in remission of manic symptoms. YMRS is an 11-item scale that measures severity of manic episodes; total score ranges from 0 (normal) to 60 (severe). Remission Rate (percent) = number of patients meeting remission criteria divided by number of patients in treatment arm, multiplied by 100.
Time Frame: 3 weeks, 6 weeks
Population: Participants in the Full Analysis Set: participants who had baseline and post-baseline measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 104 | 20 | 97
percentage of participants
  3-Week Remission Rate | 47.1 | 65.0 | 41.2
  6-Week Remission Rate | 63.5 | 60.0 | 52.6
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.384, Cochran-Mantel-Haenszel — P-value for 3-Week Remission Rate; Least Squares Mean Difference = 5.9, 95% CI 2-sided [-7.3 to 19.2] — Least Squares Mean Difference = Olanzapine minus Placebo
Statistical Analysis 2: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.982, Cochran-Mantel-Haenszel — P-value is for 6-Week Remission Rate; Least Squares Mean Difference = 0.3, 95% CI 2-sided [-21.3 to 21.8] — Least Squares Mean Difference = Olanzapine minus Haloperidol

8. Secondary Outcome: Percentage of Participants Who Switched to Symptomatic Depression
Description: Switch to symptomatic depression was defined as HAMD-17 total score ≥13 at any time in the participants with HAMD-17 total scores ≤7 at baseline. The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (normal) to 52 (severe).
Time Frame: 3 weeks, 6 weeks
Population: Participants in the Full Analysis Set (participants who had baseline and post-baseline measurement) who had HAMD-17 total scores ≤7 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 83 | 18 | 75
percentage of participants
  3-Week Symptomatic Depression Rate | 2.4 | 16.7 | 1.3
  6-Week Symptomatic Depression Rate | 2.4 | 16.7 | 2.7
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.698, Cochran-Mantel-Haenszel — P-value for 3-Week Symptomatic Depression Rate; Mean Difference (Net) = 0.8, 95% CI 2-sided [-3.2 to 4.9]
Statistical Analysis 2: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel — P-value for 6-Week Symptomatic Depression Rate; Mean Difference (Net) = -14.1, 95% CI 2-sided [-31.7 to 3.4]

9. Secondary Outcome: Change From Baseline to 3 Week and 6 Week Endpoints in the Positive Subscore of Positive and Negative Syndrome Scale (PANSS)
Description: Assesses positive symptoms associated with schizophrenia. 7 items make up the Positive scale (ex. delusions, conceptual disorganization, and hallucinatory behavior). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total Positive Subscale scores range from 7 to 49. For this study, the score was converted to 0 to 6 for each item range; hence, the total positive subscale score ranges from 0 to 42.
Time Frame: Baseline, 3 weeks, 6 weeks
Population: Participants in the Full Analysis Set: participants who had baseline and post-baseline measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 104 | 20 | 97
units on a scale
  3-Week Change | -1.8 (4.1) | -1.8 (4.3) | -0.0 (5.3)
  6-Week Change | -2.2 (4.4) | -1.6 (4.3) | -0.3 (5.7)
Statistical Analysis 1: Comparison: Olanzapine vs Placebo; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value for 3-Week Change; Least Squares Mean Difference = -1.48, 95% CI 2-sided [-2.71 to -0.25] — Least Squares Mean Difference = Olanzapine minus Placebo
Statistical Analysis 2: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.855, ANCOVA — P-value for 6-Week Change; Least Squares Mean Difference = -0.16, 95% CI 2-sided [-1.95 to 1.62] — Least Squares Mean Difference = Olanzapine minus Haloperidol

10. Secondary Outcome: Percentage of Participants Who Switched to Syndromic Depression
Description: Switch to syndromic depression was operationally defined by meeting both of the following criteria: At baseline, the symptoms did not meet the criteria for a mixed episode based on the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR). The critiera were met for a Major Depressive Episode (MDE), at any point after randomization, based on DSM-IV-TR. Rather than the 2-week period required for an MDE in the DSM-IV-TR, the patient had to meet the criteria of an MDE for at least 7 consecutive days (during Weeks 1 through 6).
Time Frame: 3 weeks, 6 weeks
Population: Participants in the Full Analysis Set (participants who had baseline and post-baseline measurement) who had manic (not mixed) episode at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 95 | 19 | 89
percentage of participants
  3-Week Syndromic Depression Rate | 0.0 | 5.3 | 0.0
  6-Week Syndromic Depression Rate | 1.1 | 5.3 | 0.0
Statistical Analysis 1: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.136, Cochran-Mantel-Haenszel — P-value for 6-Week Syndromic Depression Rate; Mean Difference (Net) = -4.6, 95% CI 2-sided [-14.9 to 5.7]

11. Secondary Outcome: Maximum Change From Baseline During 6-Week Period in Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS) Total Score
Description: Drug Induced Extra-Pyramidal Symptoms Scale (DIEPSS) is a scale used to evaluate the severity of drug induced extra-pyramidal symptoms occurring during antipsychotic drug treatment. Scale consists of 8 individual symptom scales with scores ranging from 0 (none/normal) to 4 (severe). The total score is the sum of the 8 item scores, for a total range of 0 (normal) to 32 (severe).
Time Frame: Baseline to 6 weeks
Population: Participants in the Safety Analysis Set (participants who had baseline and post-baseline measurements). Participants were included in the treatment group for which they actually received treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Haloperidol | Placebo
Number analyzed (Participants) | 105 | 20 | 96
units on a scale
  Baseline | 0.20 (0.66) | 0.50 (1.19) | 0.30 (0.91)
  Maximum Change from Baseline | 0.70 (1.51) | 2.70 (2.89) | 0.09 (1.09)
Statistical Analysis 1: Comparison: Olanzapine vs Haloperidol; Test type: Superiority or Other; p = 0.003, Wilcoxon Rank Sum — P-value for Maximum Change from Baseline

ADVERSE EVENTS:
Arm/Group | Olanzapine | Haloperidol | Placebo
Serious Adverse Events (participants affected / at risk) | 1/105 | 0/20 | 3/96
Other Adverse Events (participants affected / at risk) | 78/105 | 14/20 | 64/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=105) | Haloperidol (N=20) | Placebo (N=96)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=105) | Haloperidol (N=20) | Placebo (N=96)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (10) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Hunger (General disorders) | 3 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 6 (6) | 2 (2) | 4 (4)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Thirst (General disorders) | 16 (16) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (9) | 2 (2) | 9 (9)
Contusion (Injury, poisoning and procedural complications) | 4 (5) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 5 (5) | 0 (0) | 2 (2)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Weight increased (Investigations) | 10 (10) | 1 (1) | 4 (4)
Increased appetite (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 3 (3) | 3 (5) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 0 (0) | 1 (2)
Dystonia (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 3 (3)
Sedation (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 25 (26) | 3 (3) | 15 (17)
Tremor (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Identified errors were corrected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days